CLINICAL TRIAL: NCT03396575
Title: BRAVO: Newly-Diagnosed Brain Stem Gliomas Treated With Adoptive Cellular Therapy During Recovery From Focal Radiotherapy Alone or Focal Radiotherapy and Dose-intensified Temozolomide (Phase I)
Brief Title: Brain Stem Gliomas Treated With Adoptive Cellular Therapy During Focal Radiotherapy Recovery Alone or With Dose-intensified Temozolomide (Phase I)
Acronym: BRAVO
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Not feasible to accrue due to competing studies
Sponsor: University of Florida (Other)
Collaborators: Accelerate Brain Cancer Cure (Other); Lyla Nsouli Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB201701296; OCR16024 (Other: University of Florida)
Record Dates: First submitted 2018-01-04; First posted 2018-01-11 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Diffuse Intrinsic Pontine Glioma (DIPG); Brain Stem Glioma
Keywords: Tumor mRNA-pulsed autologous Dendritic Cells (TTRNA-DCs); Tumor-specific autologous lymphocyte transfer (TTRNA-xALT); Autologous G-CSF mobilized HSCs; Temozolomide (TMZ); Cyclophosphamide (CTX); Fludarabine (Flu); Immunotherapy; Pediatric; Young Adult; Brain Tumor; CNS; Vaccine Therapy
MeSH Terms: conditions — Diffuse Intrinsic Pontine Glioma; Xanthomatosis, Cerebrotendinous; Influenza, Human; Brain Neoplasms | interventions — Granulocyte-Macrophage Colony-Stimulating Factor; Cyclophosphamide; Diphtheria-Tetanus Vaccine

STUDY DESIGN:
Intervention Model Description: Patients in this study will either receive concurrent TMZ during RT and dose-intensive TMZ as maintenance treatment (Group A) or radiotherapy only prior to DC vaccination and without maintenance DI TMZ (Group B). Immune responses during cycles of DC vaccination with or without DI TMZ will be evaluated in both treatment groups.
  Once Group A accrual is completed and evaluated for toxicity, 6 Group B patients will be enrolled and treated at the Maximally Achievable Dose (MAD) or (Maximum Tolerated Dose) MTD determined in Group A cohort.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): TTRNA-DC vaccines with GM-CSF and TTRNA-xALT plus Td vaccine with Autologous Hematopoietic Stem cells (HSCs) during cycles of Dose-intensified TMZ
  Interventions: Biological: TTRNA-DC vaccines with GM-CSF; Biological: TTRNA-xALT; Drug: Dose-Intensified TMZ; Drug: Td vaccine; Biological: Autologous Hematopoietic Stem Cells (HSC)
- Group B (Experimental): TTRNA-DC vaccines with GM-CSF and TTRNA-xALT plus Td vaccine with Autologous Hematopoietic Stem cells (HSCs) with Cyclophosphamide + Fludarabine Lymphodepletive Conditioning
  Interventions: Biological: TTRNA-DC vaccines with GM-CSF; Biological: TTRNA-xALT; Drug: Cyclophosphamide + Fludarabine Lymphodepletive Conditioning; Drug: Td vaccine; Biological: Autologous Hematopoietic Stem Cells (HSC)

INTERVENTIONS:
Biological: TTRNA-DC vaccines with GM-CSF — After chemoradiation subjects will receive the first cycle of dose-intensified TMZ followed by three biweekly TTRNA-DC vaccines with GM-CSF. Monthly DC vaccines will be given during TMZ Cycles 2-5 for Groups A and B and 48-96 hours after completion of TMZ Cycle 6 Day 21 for Group A and 12-36 hours after HSCs for Group B. All subjects will receive an additional two bi-weekly vaccines during Cycle 6 for a total of 10 DC vaccines. All DC vaccines will be embedded with GM-CSF (150 µg per injection) and given intradermal.
Biological: TTRNA-xALT — During TMZ Cycle 4 and with DC vaccine #6, an infusion of T-cells will be administered to all subjects.
Drug: Cyclophosphamide + Fludarabine Lymphodepletive Conditioning — Subjects in Group B, however, will receive lymphodepletion with cyclophosphamide + fludarabine after DC vaccination and prior to the intravenous infusion of ex vivo expanded tumor-reactive lymphocytes.
  Arms: Group B
Drug: Dose-Intensified TMZ — After chemoradiation, subjects in Group A will receive the first cycle of dose-intensified TMZ followed by three biweekly TTRNA-DC vaccines with GM-CSF. All subjects will have an additional five cycles of dose-intensified TMZ (for a total of 6 Cycles) with concurrent monthly DC vaccinations.
  Arms: Group A
Drug: Td vaccine — A full Td booster vaccine will be administered IM at Vaccine #1 to all subjects, and vaccine site pretreatment will be administered to all subjects prior to Vaccine#3, #6, and #8.
Biological: Autologous Hematopoietic Stem Cells (HSC) — During Cycle 4, all patients will receive HSCs prior to xALT infusion and DC vaccine #6.

SUMMARY:
The standard of care for children with DIPG includes focal radiotherapy (RT) but outcomes have remained dismal despite this treatment. The addition of oral Temozolomide (TMZ) concurrently with RT followed by monthly TMZ was also found to be safe but ineffective. Recent studies in adults have shown that certain types of chemotherapy induce a profound but transient lymphopenia (low blood lymphocytes) and vaccinating and/or the adoptive transfer of tumor-specific lymphocytes into the cancer patient during this lymphopenic state leads to dramatic T cell expansion and potent immunologic and clinical responses. Therefore, patients in this study will either receive concurrent TMZ during RT and immunotherapy during and after maintenance cycles of dose-intensive TMZ (Group A) or focal radiotherapy alone and immunotherapy without maintenance DI TMZ (Group B). Immune responses during cycles of DC vaccination with or without DI TMZ will be evaluated in both treatment groups.

DETAILED DESCRIPTION:
The standard of care for children with DIPG includes external beam focal radiotherapy (RT) but outcomes have remained dismal despite this treatment. The addition of oral Temozolomide (TMZ) concurrently with focal irradiation followed by maintenance monthly TMZ was also found to be safe but ineffective. However, in the context of an immunotherapy strategy, it might be beneficial to use TMZ as an adjuvant therapy during and following radiotherapy. Recent pre-clinical and clinical studies in adults with have shown that both myeloablative (MA) and non-myeloablative (NMA) chemotherapy induce a profound but transient lymphopenia and, somewhat counterintuitively, vaccination during recovery from this lymphopenic state and/or the adoptive transfer of tumor-specific lymphocytes into lymphodepleted hosts leads to dramatic in vivo T cell expansion and potent immunologic and clinical responses. Therefore, the study team expects that tumor-specific lymphocytes, expanded ex vivo with the use of TTRNA-pulsed DCs may provide a source of lymphocytes that preferentially expand in this lymphopenic environment following TMZ, and serve as a source of responder cells to subsequent DC vaccination.

TMZ induces profound lymphopenia in children with central nervous system (CNS) tumors. It has not been conclusively shown to help in augmenting vaccine-induced immune responses in this population. Patients in this study will either receive concurrent TMZ during RT and immunotherapy during and after maintenance cycles of dose-intensive TMZ (Group A) or focal radiotherapy alone and immunotherapy without maintenance DI TMZ (Group B). Immune responses during cycles of DC vaccination with or without DI TMZ will be evaluated in both treatment groups. The immunotherapy regimen will consist of TTRNA-DC vaccines alone followed by adoptive cellular therapy consisting of ex vivo expanded tumor-reactive lymphocytes coupled with TTRNA-DC vaccines and autologous HSCs.

Patients in Group B will not receive DI TMZ, however, they will receive lymphodepletion with cyclophosphamide + fludarabine after DC vaccination and prior to the intravenous infusion of ex vivo expanded tumor-reactive lymphocytes. T cell engraftment and persistence has been shown to be augmented by lymphodepletion in numerous studies. TTRNA-pulsed DCs will be given in conjunction with the adjuvants GM-CSF and tetanus-diphtheria toxoid (Td) vaccine which the study team have shown can significantly enhance clinical responses to DC vaccination.

ELIGIBILITY:
Inclusion Criteria:

Initial Screening

* Radiologically confirmed DIPG or other diffuse intrinsic brain stem glioma (Grade III or IV).
* Patient and/or parents/guardian willing to consent to biopsy for obtaining tumor material for confirmatory diagnosis and/or tumor RNA extraction and amplification.
* Biopsy confirmation of any grade of glioma (for patients with classic DIPG on neuroimaging or at least grade III glioma in case of other diffuse intrinsic brain stem gliomas)
* Karnofsky Performance Status (KPS) of > 50% (KPS for > 16 years of age) or Lansky performance Score (LPS) of ≥ 50 (LPS for ≤ 16 years of age) assessed within 2 weeks prior to registration;
* Bone Marrow;
* ANC (absolute neutrophil count) ≥ 1000/µl (unsupported)
* Platelets ≥ 100,000/µl (unsupported)
* Hemoglobin > 8 g/dL (can be transfused)
* Renal;
* Serum creatinine ≤ upper limit of institutional normal
* Hepatic;
* Bilirubin ≤ 1.5 times upper limit of institutional normal for age
* SGPT (ALT) ≤ 3 times upper limit of institutional normal for age
* SGOT (AST) ≤ 3 times upper limit of institutional normal for age
* Patients of childbearing or child-fathering potential must be willing to use medically acceptable forms of birth control while being treated on this study.
* Signed informed consent according to institutional guidelines.

Post Biopsy

* Patients with post-surgical neurological deficits should have deficits that are stable for a minimum of 1 week prior to registration;
* Pathologic diagnosis of glioma on tumor biopsy.

Exclusion Criteria:

* Patients with severe dysphagia, obtundation, or tetraplegia (poor risks for anesthesia and biopsy procedure);
* Absence of tumor on biopsy specimen;
* Pregnant or need to breast feed during the study period (Negative serum pregnancy test required)
* Known autoimmune or immunosuppressive disease or human immunodeficiency virus infection;
* Patients with significant renal, cardiac, pulmonary, hepatic or other organ dysfunction;
* Severe or unstable concurrent medical conditions;
* Patients who require corticosteroids above physiologic doses (>4 mg/day dexamethasone) after chemoradiotherapy;
* Patients scheduled to receive any other concurrent anticancer or investigational drug therapy;
* Prior allergic reaction to TMZ, GM-CSF, or Td;
* Patients who are unwilling or unable to receive treatment and undergo follow-up evaluations at University of Florida;
* Patient and/or parent/guardian demonstrating an inability to comply with the study and/or follow-up procedures.

Ages: 3 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2018-07-17 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2025-03-20 (Actual)

PRIMARY OUTCOMES:
Feasibility and safety of adoptive cellular therapy in pediatric patients with DIPG with or without dose-intensified TMZ during cycles of DC vaccination | From first DC Vaccine through 30 days after administration of the last dose of trial drug or subject death
  Number of subjects with immunotherapy-related dose-limiting toxicities including 1) Grade III or greater non-neurologic toxicity; 2) Grade III neurologic toxicity that does not improve to Grade II or better within 5 days; or 3) Grade IV neurologic toxicity.
Determine the maximally achievable dose (MAD) or maximum tolerated dose (MTD) of xALT plus DC and HSC in Group A and Group B subjects | From first DC vaccine in Group A until 14 days after administration of the last dose of investigational product is given.
  The first 6 patients in Group A (receiving DI TMZ) at a dose of 3 x 107 cells /kg xALT and if dose-limiting toxicities are observed in no more than 1 of 6 patients, the study team will enroll another 6 patients at the next dose level of 3 x108 cells /kg. If no more than 1 patient suffers dose limiting toxicity (DLT) at this dose level, it will declared the MAD of T cells. Subjects enrolled in Group B will be treated at the MAD or MTD determined in the Group A Cohort.

SECONDARY OUTCOMES:
Post-immunotherapy functional anti-tumor immune responses | Up to 10 months
  The in vivo expansion, persistence, and function of tumor-specific lymphocytes will be followed serially in these patients using T-cell receptor (TCR) sequencing and functional immunologic analysis.
Analysis of progression-free survival (PFS) | Up to 5 years
  Days of PFS
Analysis of overall survival (OS) | Up to 5 years
  Days of OS

CONTACTS AND LOCATIONS:
Overall Officials: Elias Sayour, MD, PhD, Principal Investigator — University of Florida
Locations (1):
- UF Health Shands Children's Hospital, Gainesville, Florida, United States